CLINICAL TRIAL: NCT06789029
Title: The Effect of Dexamethasone Administration Route and Local Anesthetic Concentration on Pain, Inflammatory Response, and Neuromonitoring in Children Undergoing Scoliosis Correction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/2025
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-01

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: scoliosis; Neuromonitoring,; erector spinae plane block; dexamethasone
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- perineural Dexamethasone (Active Comparator): Erector Spinae Plane Block with 0.2% ropivacaine with perineural 0.1mg/kg dexamethasne
  Interventions: Drug: perineural Dexamethasone
- intravenous dexamethasne (Active Comparator): Erector Spinae Plane Block with 0.2% ropivacaine with intravenous 0.1mg/kg dexamethasne
  Interventions: Drug: intravenous Dexamethasone

INTERVENTIONS:
Drug: perineural Dexamethasone — Erector Spinae Plane Block with 0.2% Ropivacaine + 0.1mg/kg perineural Dexamethasone
  Arms: perineural Dexamethasone
Drug: intravenous Dexamethasone — Erector Spinae Plane Block with 0.2% Ropivacaine + 0.1mg/kg intravenous Dexamethasone
  Arms: intravenous dexamethasne

SUMMARY:
Scoliosis correction surgery in children is a complex procedure with significant risks, including postoperative pain, inflammatory response, and potential neurological complications. Effective pain control and minimizing inflammation are critical for faster recovery and improved patient outcomes. Dexamethasone is commonly used as an adjuvant in regional anesthesia due to its anti-inflammatory effects and ability to prolong analgesia. However, limited research exists on the optimal route of dexamethasone administration (intravenous vs. perineural) and the best local anesthetic concentration for pain management, inflammatory response, and neuromonitoring during surgery.

This study aims to compare the effects of different dexamethasone administration routes and local anesthetic concentrations on postoperative pain, inflammation (NLR, PLR), and neuromonitoring in pediatric scoliosis surgery. Results may improve regional anesthesia protocols, enhance patient safety, and offer valuable insights for clinical practice.

DETAILED DESCRIPTION:
Scoliosis correction surgery in children is a complex procedure associated with a significant risk of postoperative pain, inflammatory response, and potential neurological complications. Ensuring optimal pain control and minimizing adverse inflammatory responses is crucial for shortening the recovery period, improving patient comfort, and reducing the risk of long-term complications. In clinical practice, dexamethasone is frequently used as an adjuvant in regional anesthesia techniques due to its anti-inflammatory properties and its potential to prolong the analgesic effect.

Although the use of dexamethasone as an adjuvant in regional anesthesia is well known, there is limited research focusing on the impact of its route of administration (local versus intravenous) and the optimal concentration of local anesthetic agents on the effectiveness of pain control, inflammatory response, and neuromonitoring parameters during surgical procedures in children. Understanding these aspects is particularly important in complex procedures such as scoliosis correction surgery, where precise neurological function monitoring is essential for patient safety.

The objective of the proposed study is to evaluate the impact of different dexamethasone administration routes (intravenous and perineural) and varying concentrations of local anesthetic agents on postoperative pain, inflammatory response (measured using NLR and PLR indices), and neuromonitoring parameters in children undergoing scoliosis correction surgery. The findings from this study may contribute to the development of more effective and safer regional anesthesia and analgesia protocols for this patient group.

Conducting this study will provide new insights into the optimization of anesthesia in pediatric spinal surgery, potentially leading to improved treatment outcomes and patient safety, as well as valuable data for clinical practice regarding the selection of anesthetic strategies.

ELIGIBILITY:
Inclusion Criteria:

* >10 and <18 years old
* scheduled for idiopathic scoliosis surgery

Exclusion Criteria:

* included infection at the site of the regional block,
* coagulation disorders,
* immunodeficiency,
* American Society of Anesthesiologists (ASA) physical status of IV or higher,
* history of regular steroid medication.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time to first rescue opioid analgesia

SECONDARY OUTCOMES:
intraoperative requirement for propofol | durring surgery
  intraoperative requirement for propofol in mg/kg
intraoperative requirement for remifentanil | durring surgery
  intraoperative requirement for remifentanil in ug/kg
MEP | durring surgery
  Motor evoced potentials durring surgery
Total opioid consumption | 48 after surgery
  Total opioid consumption in milliequivalents of morphine per kg
NRS | 6 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 12 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 24 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 36 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NRS | 48 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
NLR | 12 hours after surgery
  Neutrophile-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophile-to-lymphocyte ratio
PLR | 12 hours after surgery
  Platelet-to-lymohocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymohocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymohocyte ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes